CLINICAL TRIAL: NCT02643550
Title: Phase 1b/2 Trial of IPH2201 And Cetuximab in Patients With Human Papillomavirus (HPV) (+) and HPV (-) Recurrent or Metastatic Squamous Cell Carcinoma of the Head and Neck
Brief Title: Study of Monalizumab and Cetuximab in Patients With Recurrent or Metastatic Squamous Cell Carcinoma of the Head and Neck
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Innate Pharma (Industry)
Collaborators: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: IPH2201-203
Record Dates: First submitted 2015-12-17; First posted 2015-12-31 (Estimated); Last update posted 2023-05-12 (Actual); Status verified 2023-05

CONDITIONS: Head and Neck Neoplasms
MeSH Terms: conditions — Head and Neck Neoplasms | interventions — monalizumab; Cetuximab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- Dose escalation (Experimental): Dose escalation of monalizumab in combination with cetuximab
  Interventions: Biological: Monalizumab; Biological: Cetuximab
- Expansion cohort 1 (Experimental): monalizumab + cetuximab expansion cohort
  Interventions: Biological: Monalizumab; Biological: Cetuximab
- Expansion cohort 2 (Experimental): monalizumab + cetuximab expansion cohort in patients with prior exposure to PD-(L)1 blockers
  Interventions: Biological: Monalizumab; Biological: Cetuximab
- Expansion cohort 3 (Experimental): monalizumab + cetuximab + anti-PD(L)1
  Interventions: Biological: Monalizumab; Biological: Cetuximab; Biological: Anti-PD(L)1

INTERVENTIONS:
Biological: Monalizumab
  Other Names: IPH2201
Biological: Cetuximab
Biological: Anti-PD(L)1
  Arms: Expansion cohort 3

SUMMARY:
The objective of this study is to evaluate in a 3 +3 design, the safety of escalating doses of Monalizumab given IV in combination with cetuximab in patients who have received prior systemic regimen(s) for recurrent and/or metastatic squamous cell carcinoma of the head and neck (SCCHN).

Cohorts expansion will evaluate antitumor activity of monalizumab and cetuximab with or without anti-PD(L)1

ELIGIBILITY:
Main Inclusion Criteria:

1. Age ≥ 18 years
2. Histologically or cytologically-confirmed, HPV (+) or HPV (-) squamous cell carcinoma of the nasopharynx (WHO Type 1), oropharynx, hypopharynx, larynx (supraglottis, glottis, subglottis) or oral cavity.
3. Recurrent or metastatic disease, documented by imaging (CT scan, MRI, X-ray) and/or physical examination with measurable disease as per Response Evaluation Criteria in Solid Tumors [RECIST] 1.1

For phase II cohorts:

* Cohort #1: Patients who received a maximum of two prior systemic regimens for recurrent and/or metastatic disease and not amenable to further therapy with curative intent
* Cohort #2: Patients with R/M SCCHN not amenable to therapy of curative intent, who have received a maximum of two prior systemic regimens in the R/M setting and who have received prior PD-(L)1 blockers
* Cohort #3: Patients with R/M SCCHN who have not received prior systemic regimens in the R/M setting and who have not received prior PD-(L)1 inhibitors

Main Exclusion Criteria:

1. For phase II cohort #1 and cohort #2: Patients who received more than 2 prior systemic regimens for recurrent and/or metastatic disease (no restriction in the phase Ib part of the trial).
2. For phase II cohort #1 and cohort #2: Patients who received cetuximab or another inhibitor of epidermal growth factor receptor are excluded from the phase II of the trial, except if cetuximab was given as part of a primary treatment approach, with no progressive disease for at least 4 months following the end of prior cetuximab treatment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 143 (Actual)
Dates: Start 2015-12; Primary Completion 2023-03-28 (Actual); Study Completion 2023-03-28 (Actual)

PRIMARY OUTCOMES:
Occurrence of Dose Limiting Toxicities (DLT) in the dose escalation part of the study | within 4 weeks after first administration
  To assess the occurrence of Drug Limited Toxicities (DLTs)
Objective Response Rate for expansion cohorts | up to 12 months
  rate of patients in complete or partial response according to RECIST 1.1.

SECONDARY OUTCOMES:
Objective Response Rate for dose escalation part of the study | up to 12 months
  rate of patients in complete or partial response according to RECIST 1.1
Duration of Response for expansion cohorts | From confirmed response until disease progression, up to 12 months
  Duration of complete and partial response
Progression Free Survival for expansion cohorts | Until disease progression or death, up to 2 years
  time between the start of treatment and the first documented progression or death
Overall Survival for expansion cohorts | Until death, up to 2 years
  time between the start of treatment and death

CONTACTS AND LOCATIONS:
Locations (18):
- United States (9):
  - University of California, Moores Cancer Center, La Jolla, California
  - Stanford Cancer Center, Stanford, California
  - University of Chicago, Chicago, Illinois
  - University of Maryland, Greenebaum Comprehensive Cancer Center, Baltimore, Maryland
  - Washington University School of Medicine, St Louis, Missouri
  - Icahn School of Medicine at Mount Sinaï, New York, New York
  - University of Pennsylvania, Philadelphia, Pennsylvania
  - Fox Chase Cancer Center, Philadelphia, Pennsylvania
  - Vanderbilt University Medical Center, Nashville, Tennessee
- France (9):
  - Centre Jean Perrin, Clermont-Ferrand
  - Centre Oscar Lambret, Lille
  - Centre Leon Berard, Lyon
  - Hopital La Timone, Marseille
  - Institut Regional du Cancer de Montpellier, Montpellier
  - Centre Antoine Lacassagne, Nice
  - Centre Eugene Marquis, Rennes
  - ICO Rene Gauducheau, Saint-Herblain
  - Institut Gustave Roussy, Villejuif

REFERENCES:
- [Derived] Hwang M, Fan C, Yue MS, Zhou D, Paturel C, Andre P, Cheng LY, Mitchell P, Kourtesis P, Ruscica D, Das M, Morsli N, Ren S, Gibbs M, Phipps A, Song X. Population Pharmacokinetics of Monalizumab in Patients With Advanced Solid Tumors. J Clin Pharmacol. 2023 Jul;63(7):817-829. doi: 10.1002/jcph.2220. Epub 2023 Apr 10. PMID 36852723